CLINICAL TRIAL: NCT05819346
Title: Effect of a Digital Lifestyle Intervention on Health-Related Quality of Life in Non-Small Cell Lung Cancer Survivors (QUALUCA): a Multicenter Randomized Controlled Trial
Brief Title: Digital Lifestyle Intervention for Lung Cancer Survivors
Acronym: QUALUCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kai-Uwe Schmitt, PhD, MEng, ICID (Other)
Responsible Party: Sponsor-Investigator, Kai-Uwe Schmitt, PhD, MEng, ICID, Sponsor, Bern University of Applied Sciences
Organization: Bern University of Applied Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Physical activity; Exercise; Nutrition; Breathing; Relaxation; Mobile application; Rehabilitation aftercare
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital lifestyle intervention (Experimental): Self-management mobile application covering physical activity, nutrition, and breathing/relaxation
  Interventions: Behavioral: Lifestyle
- Control (No Intervention): Usual care (study participation does not interfere with or change any other planned treatments)

INTERVENTIONS:
Behavioral: Lifestyle — Participants assigned to the intervention group receive access to a lifestyle mobile application for three months after rehabilitation or treatment has finished. The digital program is target group-specific and includes personalization and interactive elements without face-to-face appointments during the intervention. One virtual appointment at the beginning of the intervention with the study staff ensures that participants familiarize themselves with the mobile application and that they are assigned to a suitable program level. The intervention is mainly based on the following behavior change technique (BCT) clusters: goals and planning, feedback and monitoring, shaping knowledge, and comparison of behavior.
  Arms: Digital lifestyle intervention

SUMMARY:
The aim of this study is to assess the efficacy of a digital lifestyle intervention in non-small cell lung cancer (NSCLC) survivors on health-related quality of life (HRQoL) over three months.

DETAILED DESCRIPTION:
Lung cancer survivors suffer from reduced physical and psychological functioning as well as decreased overall health-related quality of life (HRQoL) due to cancer symptoms, cancer treatments, and comorbidities. Experienced symptoms by lung cancer survivors, such as cancer-related fatigue or dyspnea, persist after active treatment ends. Therefore, lung cancer survivors should receive continuous attention regarding their health and HRQoL beyond the expected cancer cure.

Physical activity, healthy nutrition, and breathing/relaxation exercises before, during, and after cancer treatments can increase physical as well as psychological functioning and HRQoL. Thus, the adhesion to an appropriate healthy lifestyle is crucial and represents an effective adjunctive strategy in the management of lung cancer survivors. Most lung cancer survivors, however, are sedentary and fail to meet official lifestyle recommendations, for instance, of the American Cancer Society or the World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR).

The present project evaluates a mobile application for non-small cell lung cancer (NSCLC) survivors that will be used for three months after rehabilitation or treatment has finished. The main foci of the mobile application are physical activity, nutrition, and breathing/relaxation. The contents of the mobile application and the mobile application itself were developed in an iterative co-creation process involving software developers and potential users as well as researchers and clinicians from different disciplines (e.g., physical therapy and nutritional therapy).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of non-small cell lung cancer (NSCLC)
* Estimated life expectancy of ≥ six months (judged by local investigators/responsible health professionals)
* Undergoing inpatient or outpatient rehabilitation OR completion of planned surgery, chemotherapy, or radiation therapy for NSCLC within the past 24 weeks
* Knowledge of German to understand study material and assessments
* Access to a cell phone or tablet
* Written informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Inability to participate in the intervention because of physical, cognitive, or safety reasons (judged by local investigators/responsible health professionals)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (Scale-Global health status) | Change from baseline to 3 months
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) (2 items; 7-point Likert-type scale; the score ranges from 0 to 100; a high score for the global health status represents a high HRQoL)

SECONDARY OUTCOMES:
Health-related quality of life (5 functional scales, 9 symptom scales/items) | Change from baseline to 3 months
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) (28 items; 4-point Likert-type scale; 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning), 3 symptom scales (fatigue, nausea and vomiting, pain), 6 single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties); all scales and single-item measures range in score from 0 to 100)
Lung cancer-specific health-related quality of life (10 symptom scales/items) | Change from baseline to 3 months
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 29 (lung cancer-specific module) (EORTC QLQ-LC29) (29 items; 4-point Likert-type scale / 5 multi-item scales and 5 single items; all scales and single-item measures range in score from 0 to 100)
Body mass index [kg/m²] | Change from baseline to 3 months
  Computed using self-reported body weight [kg] and height [m]
Physical activity (self-reported) | Change from baseline to 3 months
  Modified Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ) (physical activity before rehabilitation/treatment and physical activity over the last week)
Functional exercise capacity | Change from baseline to 3 months
  1-Minute Sit-to-Stand Test (number of repetitions)
Risk for low protein intake | Change from baseline to 3 months
  Protein Screener 55+ (Pro55+) (10 items)
Appetite | Change from baseline to 3 months
  Simplified Nutritional Appetite Questionnaire (SNAQ) (4 items; 5-point Likert-type scale)
Psychological distress | Change from baseline to 3 months
  Short form of the Patient Health Questionnaire (PHQ-4) (4 items)
Cancer-related fatigue | Change from baseline to 3 months
  Brief Fatigue Inventory (BFI) (9 items)
Enablement | Change from baseline to 3 months
  Shortened version of the Patient Enablement Scale-13 (PEN-13) (5 out of 13 items; 5-point Likert-type scale)
Self-rated health | Weekly for 3 months
  EuroQol Group Visual Analogue Scale (EQ VAS) (vertical visual analog scale that takes values between 100 [best imaginable health] and 0 [worst imaginable health], on which respondents provide a global assessment of their health)

OTHER OUTCOMES:
Usability (intervention group only) | At 3 months follow-up (end of the intervention)
  mHealth App Usability Questionnaire (MAUQ)
Acceptability, appropriateness, and feasibility (intervention group only) | At 3 months follow-up (end of the intervention)
  Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) (4-item measures of implementation outcomes)
Experiences and satisfaction with the digital lifestyle intervention (intervention group only) | At 3 months follow-up (end of the intervention)
  Short semi-structured interview; outcomes will be qualitatively assessed (no scale is used)
Treatments/support since baseline | At 3 months follow-up (end of the intervention)
  Cancer treatments (e.g., chemotherapy) and therapies/support (e.g., physical therapy, self-help group) participants might have received during the last 3 months (2 items)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Frei, PhD, Principal Investigator — University of Zurich
Locations (4):
- Switzerland (4):
  - Klinik Barmelweid AG, Barmelweid
  - Zürcher RehaZentren | Klinik Davos, Davos
  - Berner Reha Zentrum AG, Heiligenschwendi
  - Zürcher RehaZentren | Klinik Wald, Wald

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized data will be made available upon reasonable request after the main results have been published. The privacy of each subject and confidentiality of their information will be preserved in reports and publication of data.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Weber M, Raab AM, Schmitt KU, Busching G, Marcin T, Spielmanns M, Puhan MA, Frei A. Efficacy of a digital lifestyle intervention on health-related QUAlity of life in non-small cell LUng CAncer survivors following inpatient rehabilitation: protocol of the QUALUCA Swiss multicentre randomised controlled trial. BMJ Open. 2024 Mar 7;14(3):e081397. doi: 10.1136/bmjopen-2023-081397. PMID 38453202